CLINICAL TRIAL: NCT07183852
Title: Locoregional or Systemic Administration of Autologous Tumor Infiltrating Lymphocytes in Patients With Metastatic Melanoma
Acronym: GoTIL-01
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GoTIL_2025EU
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Uveal Melanoma; Metastatic Cutaneous Melanoma
Keywords: Adoptive Cell Therapy; Tumor Infiltrating Lymphocyte; Hepatic Arterial Infusion; Melphalan; Interleukin-2
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Melphalan; Interleukin-2

STUDY DESIGN:
Intervention Model Description: Cohort 1 Patients With Uveal Melanoma and Liver Metastases, locoregional admin using HAI
  Cohort 2 Patients With Cutaneous Melanoma and visceral metastases, IV admin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients With Uveal Melanoma and Liver Metastases, locoregional admin using HAI
  Interventions: Drug: Autologous Tumor Infiltrating Lymphocytes (TIL); Drug: Melphalan; Drug: Interleukin-2
- Cohort 2 (Experimental): Patients With Cutaneous Melanoma and visceral metastases, IV admin
  Interventions: Drug: Autologous Tumor Infiltrating Lymphocytes (TIL); Drug: Melphalan; Drug: Interleukin-2

INTERVENTIONS:
Drug: Autologous Tumor Infiltrating Lymphocytes (TIL) — Cohort 1: Administered via hepatic arterial infusion Cohort 2: Administered via intravenous infusion
Drug: Melphalan — 1 mg/kg, IV
Drug: Interleukin-2 — 2 MIU, subcutaneous twice daily for up to 14 days.

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety and tolerability of locoregional or systemic administration of autologous tumor infiltrating lymphocytes in patients with metastatic melanoma

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 18 years of age.
2. Can provide a signed informed consent as described in the protocol, including compliance with the requirements and restrictions listed in the ICF and in this protocol.
3. World Health Organization (WHO) Performance Status 0 or 1.
4. Patient must have a histologically/cytologically confirmed diagnosis of:

   * stage IV uveal melanoma with confirmed progression following prior systemic therapy with tebentafusp (if HLA A2:01 positive) OR
   * stage IV cutaneous melanoma with confirmed progression following prior systemic therapy with a programmed cell death protein-1 (PD-1) inhibitor with or without a CTLA-4 inhibitor
5. At least one resectable lesion in the liver (or aggregate of lesions resected) of a minimum size of 0.5 cm in diameter to generate TILs.
6. Measurable disease by computed tomography (CT) per RECIST 1.1 criteria after resection of lesion for TILs production
7. No other malignancies, except if treated with curative intent and with a cancer-related life expectancy of more than 5 years.
8. Female patient of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female patients of childbearing potential must be willing to use a highly efficient method of contraception (Pearl index <1), for the course of the study through 120 days after the last dose of study medication.
10. Male patients with women of childbearing potential partners must agree to use a condom for contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Any serious or uncontrolled medical conditions that, in the investigator's opinion, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy (including operation), or interfere with the interpretation of study results.
2. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
3. Women who are pregnant or breastfeeding.
4. Any condition that potentially hamper compliance with the study protocol and follow-up schedule; those conditions should be discussed with the subject before registration in the trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 5 years
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs). graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  RECIST 1.1
Progression free-survival (PFS) | 2 years
  Evaluation of Progression-free survival
hepatic Progression-free survival (hPFS) | 2 years
  Evaluation of hepatic Progression-free survival
Duration of objective response (DOR) | 2 years
  Evaluation of duration of a response by RECIST 1.1
Overall Survival (OS) | 5 years
  Evaluation of Overall Survival
Evaluation of feasibility of an automated production of TILs | 2 years
  Defined as the proportion of patients included that receive treatment with the TIL product.

IPD SHARING:
Plan to Share IPD: Undecided